CLINICAL TRIAL: NCT02375854
Title: Outcomes of Neonatal Acute Kidney Injury and Prematurity: An Observational Study and Einstein-Montefiore Neonatal Acute Kidney Injury Clinical Registry and Biorepository
Brief Title: Outcomes of Neonatal Acute Kidney Injury In Premature Infants
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-2900
Record Dates: First submitted 2015-02-19; First posted 2015-03-03 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Kidney Injury; Chronic Kidney Disease
Keywords: preterm; acute kidney injury; biomarkers; chronic kidney disease
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic; Premature Birth | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infants: Less than 32 weeks' gestation
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
The objective of this protocol is to investigate the impact of prematurity, with or without associated acute kidney injury (AKI), on the future risk of chronic kidney disease (CKD) by establishing a patient registry and biorepository. Serum and urine samples will be collected serially from premature infants admitted to the neonatal intensive care unit (NICU) at Albert Einstein College of Medicine/Weiler Hospital and subsequently followed in the NICU follow-up and pediatric nephrology ambulatory subspecialty clinics. The biorepository will be linked to a comprehensive clinical database.

DETAILED DESCRIPTION:
This is an observational pilot study to enhance understanding of the pathophysiology and epidemiology associated with effects of AKI in premature infants and the role that neonatal AKI plays in future development of CKD. In eligible preterm infants, blood and urine samples will be collected at pre-specified time points during hospitalization and at outpatient follow-up appointments at 6 months, 1 year, 2 years, and 5 years of age and stored in the biorepository. Blood pressure will be measured and recorded at NICU discharge and at all follow-up visits. A renal ultrasound will be performed to monitor renal growth at 2 and 5 years of age. All data will be entered into a comprehensive clinical database, including laboratory results.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 32 weeks/ gestational age admitted to the Neonatal Intensive Care Unit at Weiler Hospital (The Children's Hospital at Montefiore).

Exclusion Criteria:

* Known major congenital anomalies of the kidney and urinary tract (CAKUT) including solitary kidney, cystic dysplasia, multicystic dysplastic kidney, renal hypoplasia, obstructive uropathy
* Other genetic syndromes or medical conditions that preclude enrollment per judgment of the attending neonatologist

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants less than 32 weeks' gestational age
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Chronic kidney disease (incidence of chronic renal insufficiency in childhood) | 5 years
  Determine the incidence of chronic renal insufficiency in childhood

SECONDARY OUTCOMES:
Acute kidney injury (incidence of acute kidney injury in preterm infants) | 0-5 months
  Determine the incidence of acute kidney injury in preterm infants
Assessment of serum biomarkers - cystatin C | 0 months - 5 years
  Determination of serum and urinary biomarkers to predict the development of acute kidney injury and chronic renal insufficiency
Assessment of urinary biomarkers - urinary neutrophil gelatinase-associated lipocalin, interlukin 18 and kidney-injury molecule-1 | 0 months - 5 years
  Determination of serum and urinary biomarkers to predict the development of acute kidney injury and chronic renal insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Fuloria, MD, Principal Investigator — The Children's Hospital at Montefiore, Albert Einstein College of Medicine
Locations (1):
- Jack D. Weiler Hospital, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No